CLINICAL TRIAL: NCT03704766
Title: Alpha-Defensin and Synovial Proteins to Improve Detection of Pediatric Septic Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other); Children's Healthcare of Atlanta (Other); Campbell Clinic (Other); CD Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015-947
Record Dates: First submitted 2018-05-08; First posted 2018-10-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-06

CONDITIONS: Joint Infection; Infection of Hip Joint (Disorder); Infection of Shoulder Joint; Septic Arthritis
Keywords: synovial biomarkers; alpha-defensin; diagnostics; pediatric
MeSH Terms: conditions — Arthritis, Infectious | interventions — Blood Cell Count; Blood Culture

STUDY DESIGN:
Intervention Model Description: Participants are assigned as either cases of infection/inflammation, or normative controls, and receive the same diagnostic testing for the duration of the study.
Who Masked: Participant, Care Provider
Masking Description: For patients with inflamed joints, the medical team will be blind to the results of the alpha-defensin assay and other experimental tests for a period of 2 weeks, after which results may be divulged to the clinical team at their request. As such, the results will not influence the physician/surgeons' decision for acute treatment of the patient, as the decision to treat suspected septic arthritis is typically made within 24 hours, and the final diagnosis is made within 2 weeks (pending culture results). As the testing of the leukocyte esterase strips will occur in the operating room, the surgeon will not be blinded to these results. A blinded team member will read the pictures of all of the leukocyte test strip results at once, after they have all been collected. The patient will be made aware of results at the physician/surgeon's discretion. For normative controls, the results of experimental testing will not be divulged to the clinical team or to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inflamed/Infected Joint (Experimental): Patients undergoing joint aspiration/debridement due to suspicion of septic joint or rheumatologic/inflammatory condition
  Interventions: Diagnostic Test: Synovial Alpha-defensin assay; Diagnostic Test: Synovial Neutrophil elastase assay; Diagnostic Test: Synovial lactate assay; Diagnostic Test: Synovial C-reactive Protein (CRP); Diagnostic Test: Synovial Staphylococcus spp antigen panel; Diagnostic Test: Synovial Candida spp antigen panel; Diagnostic Test: Synovial Enterococcus faecalis assay; Diagnostic Test: Synovial bacterial culture by BacT/Alert; Diagnostic Test: Synovial Cell count + differential (CBC); Diagnostic Test: Synovial Gram Stain; Diagnostic Test: Synovial Leukocyte Esterase Test Strips; Diagnostic Test: Synovial PCR for Kingella kingae; Diagnostic Test: Serum Cell count + differential (CBC); Diagnostic Test: Serum erythrocyte sedimentation rate (ESR); Diagnostic Test: Serum C-reactive Protein (CRP); Diagnostic Test: Serum D-dimer; Diagnostic Test: Serum Procalcitonin; Diagnostic Test: Blood Cultures; Diagnostic Test: Optional blood testing per standard of care (ASO, anti-strep, ANA, anti-DS-DNA, HLA-B27, RF, Lyme and other inflammatory/ rheumatologic markers )
- Normative Control (Active Comparator): Patient undergoing procedure unrelated to infection/inflammation
  Interventions: Diagnostic Test: Synovial Alpha-defensin assay; Diagnostic Test: Synovial Neutrophil elastase assay; Diagnostic Test: Synovial lactate assay; Diagnostic Test: Synovial C-reactive Protein (CRP); Diagnostic Test: Synovial Staphylococcus spp antigen panel; Diagnostic Test: Synovial Candida spp antigen panel; Diagnostic Test: Synovial Enterococcus faecalis assay; Diagnostic Test: Synovial bacterial culture by BacT/Alert; Diagnostic Test: Synovial Cell count + differential (CBC); Diagnostic Test: Synovial Gram Stain; Diagnostic Test: Synovial Leukocyte Esterase Test Strips; Diagnostic Test: Synovial PCR for Kingella kingae; Diagnostic Test: Serum Cell count + differential (CBC); Diagnostic Test: Serum erythrocyte sedimentation rate (ESR); Diagnostic Test: Serum C-reactive Protein (CRP); Diagnostic Test: Serum D-dimer; Diagnostic Test: Serum Procalcitonin; Diagnostic Test: Blood Cultures; Diagnostic Test: Optional blood testing per standard of care (ASO, anti-strep, ANA, anti-DS-DNA, HLA-B27, RF, Lyme and other inflammatory/ rheumatologic markers )

INTERVENTIONS:
Diagnostic Test: Synovial Alpha-defensin assay — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial Neutrophil elastase assay — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial lactate assay — Synovial Fluid (joint fluid) will be sent out to CD Diagnostics for this test.
Diagnostic Test: Synovial C-reactive Protein (CRP) — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial Staphylococcus spp antigen panel — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial Candida spp antigen panel — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial Enterococcus faecalis assay — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial bacterial culture by BacT/Alert — The synovial fluid (joint fluid) sent to CD Diagnostics for testing will also be cultured to see if any organisms grow.
Diagnostic Test: Synovial Cell count + differential (CBC) — One of the synovial fluid (joint fluid) tests that will be performed by the outside lab, CD Diagnostics.
Diagnostic Test: Synovial Gram Stain — This will be performed by CD Diagnostics if any organisms are present in the synovial fluid.
Diagnostic Test: Synovial Leukocyte Esterase Test Strips — These test strips will be tested at the hospital where the patient is being seen, a few drops of synovial fluid will be used on the strip.
Diagnostic Test: Synovial PCR for Kingella kingae — In participants < 8 years old, a sample of synovial fluid will be tested for Kingella kingae using PCR.
Diagnostic Test: Serum Cell count + differential (CBC) — A blood test performed at the hospital.
Diagnostic Test: Serum erythrocyte sedimentation rate (ESR) — A blood test performed at the hospital.
Diagnostic Test: Serum C-reactive Protein (CRP) — A blood test performed at the hospital.
Diagnostic Test: Serum D-dimer — A blood test performed at the hospital.
Diagnostic Test: Serum Procalcitonin — A blood test performed at the hospital.
Diagnostic Test: Blood Cultures — Blood will be cultured at the hospital to see if any organisms grow.
Diagnostic Test: Optional blood testing per standard of care (ASO, anti-strep, ANA, anti-DS-DNA, HLA-B27, RF, Lyme and other inflammatory/ rheumatologic markers ) — In patients with suspected inflammation/infection, there are other blood tests which may be standard of care and used for diagnosis.

SUMMARY:
Differentiating between septic arthritis and other causes of joint inflammation in pediatric patients is challenging and of the utmost importance because septic arthritis requires surgical debridement as part of the treatment regimen. The current gold standard to diagnose septic arthritis in children is a positive synovial fluid culture; however, joint cultures may take several days to return. If a bacterial infection is present, it requires immediate surgical intervention in order to prevent lasting articular cartilage damage. Frequently surgeons must decide whether to surgically debride a joint before culture results are available. There is no single lab test or clinical feature that reliably indicates bacterial infection over other causes of joint inflammation. The alpha-defensin assay has shown high sensitivity and specificity for joint infection in other studies.The purpose of this study is to determine the sensitivity and specificity of several synovial biomarkers for diagnosing pediatric septic arthritis.

DETAILED DESCRIPTION:
The purpose of this study is to determine if alpha-defensin and other proteins present in joint fluid may be able to rapidly diagnose bacterial joint infections. Patients with suspected joint infection typically undergo joint aspiration so that tests can be performed to help diagnose joint infection, including gram stain, cell count, and culture. Patients under 18 years old that are undergoing sampling of their joint fluid due to suspicion of infection or inflammation will be enrolled in this multi-center trial. Joint fluid will also be sampled from normative controls made up of patients who are undergoing an unrelated procedure without inflammation or infection. Joint fluid from patients with suspected inflammation/infection and from normative controls will be analysed for presence of alpha-defensin, leukocyte esterase, neutrophil elastase, synovial C-reactive protein, and synovial lactate. The alpha-defensin assay has shown high sensitivity and specificity for joint infection in other studies. Additionally a Staphylococcus spp antigen panel, Candida spp antigen panel, Enterococcus faecalis assay, BACTAlert culture, cell count plus differential, gram stain, and aerobic, anaerobic, and fungal cultures will be done using synovial fluid. A synovial fluid PCR for Kingella kingae will be performed if the patient is under eight years of age. Blood tests will include cell count and differential, erythrocyte sedimentation rate, C-reactive protein, procalcitonin, and D-dimer, as well as relevant inflammatory or rheumatologic marker tests. Results from these tests will be compared to joint fluid culture which the gold standard for diagnosing bacterial infection. The study includes 1 visit per patient, the standard of care visit in which the patient would be undergoing joint aspiration or arthroscopy. Once data has been collected, the sensitivity and specificity will be determined for these experimental tests both individually and in combination.

ELIGIBILITY:
Inclusion Criteria- Septic Cases and Inflamed, Non-Septic Comparators:

* Synovial fluid is obtained to assess for infection or inflammatory/rheumatologic disease (all medium and large joints will be included: hip, knee, ankle, shoulder, subtalar, elbow, and wrist joints)
* Patients with recent antibiotic exposure are eligible to participate but will be analyzed separately

Inclusion Criteria- Normative Controls:

* Patients undergoing a procedure unrelated to infection (the procedure may be arthroscopy, or an open or percutaneous bony or soft tissue procedure)

Exclusion Criteria- All Participants:

* Family declines to participate/consent
* Patients with a major joint trauma (such as a documented ligament tear or fracture) within the past 8 weeks are not eligible to have that joint aspirated, but could have another joint aspirated

Exclusion Criteria- Normative Controls:

* A history of recent infection (within the past 3 months)
* Received antibiotics in the past 7 days

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 442 (Estimated)
Dates: Start 2016-06-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of experimental tests | Interim analysis at 2 years of study recruitment
  Sensitivity and specificity have been selected as these are standard outcome tests when determining the utility of a diagnostic test.

CONTACTS AND LOCATIONS:
Overall Officials: Emily R Dodwell, MD, MPH, Principal Investigator — The Hospital for Special Surgery
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Hospital for Special Surgery, New York, New York
  - Campbell Clinic, Collierville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Collaborating sites will share de-identified patient data with the primary site, the Hospital for Special Surgery. The Hospital for Special Surgery, will incorporate de-identified aggregated data into a separate de-identified aggregated data sat to be provided to all study sites, but individual participant data will not be shared with all sites.

REFERENCES:
- [Background] Bingham J, Clarke H, Spangehl M, Schwartz A, Beauchamp C, Goldberg B. The alpha defensin-1 biomarker assay can be used to evaluate the potentially infected total joint arthroplasty. Clin Orthop Relat Res. 2014 Dec;472(12):4006-9. doi: 10.1007/s11999-014-3900-7. Epub 2014 Sep 26. PMID 25256621
- [Background] Brook I, Reza MJ, Bricknell KS, Bluestone R, Finegold SM. Synovial fluid lactic acid. A diagnostic aid in septic arthritis. Arthritis Rheum. 1978 Sep-Oct;21(7):774-9. doi: 10.1002/art.1780210706. PMID 697948
- [Background] Carpenter CR, Schuur JD, Everett WW, Pines JM. Evidence-based diagnostics: adult septic arthritis. Acad Emerg Med. 2011 Aug;18(8):781-96. doi: 10.1111/j.1553-2712.2011.01121.x. PMID 21843213
- [Background] Colvin OC, Kransdorf MJ, Roberts CC, Chivers FS, Lorans R, Beauchamp CP, Schwartz AJ. Leukocyte esterase analysis in the diagnosis of joint infection: can we make a diagnosis using a simple urine dipstick? Skeletal Radiol. 2015 May;44(5):673-7. doi: 10.1007/s00256-015-2097-5. Epub 2015 Jan 29. PMID 25626524
- [Background] Cunningham G, Seghrouchni K, Ruffieux E, Vaudaux P, Gayet-Ageron A, Cherkaoui A, Godinho E, Lew D, Hoffmeyer P, Uckay I. Gram and acridine orange staining for diagnosis of septic arthritis in different patient populations. Int Orthop. 2014 Jun;38(6):1283-90. doi: 10.1007/s00264-014-2284-3. Epub 2014 Feb 5. PMID 24496757
- [Background] Deirmengian C, Kardos K, Kilmartin P, Cameron A, Schiller K, Parvizi J. Combined measurement of synovial fluid alpha-Defensin and C-reactive protein levels: highly accurate for diagnosing periprosthetic joint infection. J Bone Joint Surg Am. 2014 Sep 3;96(17):1439-45. doi: 10.2106/JBJS.M.01316. PMID 25187582
- [Background] Deirmengian C, Kardos K, Kilmartin P, Gulati S, Citrano P, Booth RE Jr. The Alpha-defensin Test for Periprosthetic Joint Infection Responds to a Wide Spectrum of Organisms. Clin Orthop Relat Res. 2015 Jul;473(7):2229-35. doi: 10.1007/s11999-015-4152-x. PMID 25631170
- [Background] Frangiamore SJ, Saleh A, Grosso MJ, Kovac MF, Higuera CA, Iannotti JP, Ricchetti ET. alpha-Defensin as a predictor of periprosthetic shoulder infection. J Shoulder Elbow Surg. 2015 Jul;24(7):1021-7. doi: 10.1016/j.jse.2014.12.021. Epub 2015 Feb 8. PMID 25672257
- [Background] Gafur OA, Copley LA, Hollmig ST, Browne RH, Thornton LA, Crawford SE. The impact of the current epidemiology of pediatric musculoskeletal infection on evaluation and treatment guidelines. J Pediatr Orthop. 2008 Oct-Nov;28(7):777-85. doi: 10.1097/BPO.0b013e318186eb4b. PMID 18812907
- [Background] Ganz T, Selsted ME, Szklarek D, Harwig SS, Daher K, Bainton DF, Lehrer RI. Defensins. Natural peptide antibiotics of human neutrophils. J Clin Invest. 1985 Oct;76(4):1427-35. doi: 10.1172/JCI112120. PMID 2997278
- [Background] Hatakeyama Y, Miura H, Sato A, Onodera Y, Sato N, Shimizu D, Kumazawa Y, Sanada H, Hirano H, Terada Y. Neutrophil elastase in amniotic fluid as a predictor of preterm birth after emergent cervical cerclage. Acta Obstet Gynecol Scand. 2016 Oct;95(10):1136-42. doi: 10.1111/aogs.12928. Epub 2016 Jun 17. PMID 27216361
- [Background] Heyworth BE, Shore BJ, Donohue KS, Miller PE, Kocher MS, Glotzbecker MP. Management of pediatric patients with synovial fluid white blood-cell counts of 25,000 to 75,000 cells/mm(3) after aspiration of the hip. J Bone Joint Surg Am. 2015 Mar 4;97(5):389-95. doi: 10.2106/JBJS.N.00443. PMID 25740029
- [Background] Maharajan K, Patro DK, Menon J, Hariharan AP, Parija SC, Poduval M, Thimmaiah S. Serum Procalcitonin is a sensitive and specific marker in the diagnosis of septic arthritis and acute osteomyelitis. J Orthop Surg Res. 2013 Jul 4;8:19. doi: 10.1186/1749-799X-8-19. PMID 23826894
- [Background] Potter BK. From Bench to Bedside: Alpha-defensing--The Biggest Thing in Joint Replacement Infections Since Prophylactic Antibiotics? Clin Orthop Relat Res. 2015 Oct;473(10):3105-7. doi: 10.1007/s11999-015-4297-7. Epub 2015 Apr 14. No abstract available. PMID 25869063
- [Background] Nakamura A, Osonoi T, Terauchi Y. Relationship between urinary sodium excretion and pioglitazone-induced edema. J Diabetes Investig. 2010 Oct 19;1(5):208-11. doi: 10.1111/j.2040-1124.2010.00046.x. PMID 24843434
- [Background] Riise OR, Kirkhus E, Handeland KS, Flato B, Reiseter T, Cvancarova M, Nakstad B, Wathne KO. Childhood osteomyelitis-incidence and differentiation from other acute onset musculoskeletal features in a population-based study. BMC Pediatr. 2008 Oct 20;8:45. doi: 10.1186/1471-2431-8-45. PMID 18937840
- [Background] Wang C, Wang Q, Li R, Duan JY, Wang CB. Synovial Fluid C-reactive Protein as a Diagnostic Marker for Periprosthetic Joint Infection: A Systematic Review and Meta-analysis. Chin Med J (Engl). 2016 Aug 20;129(16):1987-93. doi: 10.4103/0366-6999.187857. PMID 27503025
- [Background] Wyatt MC, Beswick AD, Kunutsor SK, Wilson MJ, Whitehouse MR, Blom AW. The Alpha-Defensin Immunoassay and Leukocyte Esterase Colorimetric Strip Test for the Diagnosis of Periprosthetic Infection: A Systematic Review and Meta-Analysis. J Bone Joint Surg Am. 2016 Jun 15;98(12):992-1000. doi: 10.2106/JBJS.15.01142. PMID 27307359
- See also: Leukocyte esterase reagent strips for the rapid diagnosis of periprosthetic joint infection — https://pubmed.ncbi.nlm.nih.gov/22608686/